CLINICAL TRIAL: NCT02984410
Title: Phase III Study Assessing the "Best of" Radiotherapy Compared to the "Best of" Surgery (Trans-oral Surgery (TOS)) in Patients With T1-T2, N0-N1 Oropharyngeal, Supraglottic Carcinoma and With T1, N0 Hypopharyngeal Carcinoma
Brief Title: Study Assessing The "Best of" Radiotherapy vs the "Best of" Surgery in Patients With Oropharyngeal Carcinoma
Acronym: Best Of
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1420-HNCG-ROG
Record Dates: First submitted 2016-11-28; First posted 2016-12-06 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Oropharyngeal Cancer; Supraglottic Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma
Keywords: T1-T2, N0-N1 oropharyngeal carcinoma, supraglottic carcinoma, T1, N0 hypopharyngeal carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensity-Modulated Radiation Therapy (IMRT) (Other): PTV prescription to tumor and high risk areas will be delivered daily for 5 days per week to a total dose of 66-70Gy in 2 Gy/fraction over 6 weeks, elective/prophylactic mucosal and nodal areas will receive a total dose of 54.25- 54.45 Gy in 33-35 fractions of 1.55-1.65 Gy over 6 weeks.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT)
- Trans Oral Surgery (TOS) (Other): The following surgical techniques are allowed:
  Transoral Robotic Surgery (TORS) Transoral Microsurgery (TLM) Conventional trans-oral Surgery (CTOS)
  Interventions: Procedure: Trans Oral Surgery (TOS)

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — IMRT (Simultaneous Integrated Boost (SIB) and accelerated regimen) with selective neck node dissection
  Arms: Intensity-Modulated Radiation Therapy (IMRT)
Procedure: Trans Oral Surgery (TOS) — TOS (Trans Oral Laser Microsurgery (TLM), Trans Oral Robotic Surgery (TORS), conventional) with selective neck node dissection
  Arms: Trans Oral Surgery (TOS)

SUMMARY:
Oropharyngeal Squamous Cell Carcinoma (OPSCC) arises in the soft palate, tonsils, base of tongue, pharyngeal wall, and the vallecula. Most of the patients with early stage OPSCC are usually cured. Treatment of early stage OPSCC can be successfully achieved with primary surgery including neck dissection, as indicated, or with definitive radiotherapy. The current standard treatment for OPSCC is therefore based on either surgery and/or radiotherapy, both associated with comparable, high tumor control rates but with different side effects profiles and technical constraints.

In order to decrease the potential morbidity of surgery, transoral approaches have been developed within the last decades, including transoral robotic surgery (TORS), transoral laser microsurgery (TLM) or conventional transoral techniques. On the other hand, patients with head and neck cancer treated with IMRT experienced significant improvements in cause specific survival (CSS) compared with patients treated with non-IMRT techniques thus suggesting that IMRT may be beneficial in terms of patient's outcomes and toxicity profile. It is as yet unclear however, which one of the new techniques is superior to the other in terms of function preservation. Given that the functional outcome of most importance is swallowing function, the preservation of swallowing is thus of major importance.

The main objective of the study is to assess and compare the patient-reported swallowing function over the first year after randomization to either IMRT or TOS among patients with early stage OPSCC, SGSCC, and HPSCC.

DETAILED DESCRIPTION:
Eligible patients will be randomized 1 to 1 to surgery (Arm 1) or radiotherapy (Arm 2).

ARM 1: Surgery

Trans-oral surgery (any trans-oral approach such as trans-oral laser microsurgery conventional trans-oral surgery or trans-oral robotic surgery) will be applied to all patients in this arm.

A surgical margin is defined to be clear (R0), if found to be >/=3mm in the final specimen (except deep margin for tonsillar resection, that is either R1 or R0), is defined to be close, if 1-<3mm, and considered to be involved (R1), if <1mm in the final specimen. Clearly defined marginal biopsies are required for each TOS-technique. Trans-oral re-resections are required in case of R1 or close-margin to convert the patient to an R0-status.Postoperative RT or chemo-RT will be given within 5-6 weeks of surgery in case of positive.

ARM 2: Radiotherapy

Intensity modulated radiation therapy (IMRT) with Simultaneous integrated boost (SIB) will be applied to all patients in this arm. PTV prescription to tumor and high risk areas will be delivered daily for 5 days per week to a total dose of 66-70Gy in 2 Gy/fraction over 6 weeks, elective/prophylactic mucosal and nodal areas will receive a total dose of 54.25- 54.45 Gy in 33-35 fractions of 1.55-1.65 Gy over 6 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

* OPSCC in one of the following sub-sites: base of tongue, lateral pharyngeal wall, tonsil, glosso-tonsillar sulcus, vallecula or SGSCC in one or more of the following sub-sites: epiglottis, aryepiglottic fold, false cord or HPSCC in one or more of the following subsites: Lateral and medial wall of piriform sinus (sub-sites are defined as lateral (lateral pharyngeal wall, tonsil, glosso-tonsillar sulcus, lateral piriform sinus) vs. central lesions (base of tongue, vallecula, all supraglottic sites, medial wall of piriform sinus))
* TNM stage I-III (7th AJCC classification): T1 or T2, N0 or T1 or T2, N1 with one single neck node ≤ 3cm without radiographic signs of extracapsular extension (ECE), M0;
* TNM stage I for HPSCC: T1, N0, M0. ;
* Within 2 weeks before randomization, assessment by a Multi-Disciplinary Team (MDT) composed of at least a head and neck/ENT surgeon, oncologist, radiologist, radiotherapist, and pathologist of the treatment naïve patient and suitable for either TOS or IMRT based on:
* CT with contrast and/or MRI done within 4 weeks prior to randomization Note: Repeat contrast enhanced CT and/or MRI or US 1 week or less prior to randomization in case of suspicious nodes <1cm on initial scan if per local practice
* Pan-endoscopy with assessment of trans-oral exposure for resection.
* peri-nodal infiltration either via CT-scan or MRI.
* Age 18 and older; Age 18 to 70 for SGSCC
* ECOG Performance status ≤ 2;
* Availability of biological material for HPV/p16 testing for OPSCCs
* Study information and Informed consent discussed by the surgeon and radio-oncologist and signed by the patient.
* Within 2 weeks prior randomization:
* Baseline MDADI score available;
* Adequate bone marrow function as demonstrated by neutrophils count > 1,5 109 /L , platelets count > 75 109 /L, WBC≥ 3.0 109 /L;
* Prothrombin time (PT) with an international normalized ratio (INR) ≤ 1.2
* Partial thromboplastin time (PTT) ≤ 1.2 times ULN
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test no more than 72 hours prior to randomization.
* Patients of childbearing / reproductive potential should agree to use adequate birth control measures for 3 months, especially if they will undergo any radiotherapy treatment at any time during the study. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

Main Exclusion Criteria:

* Any previous anti-cancer therapy for HNSCC (surgery, chemo-, or radiotherapy or molecular targeted therapy);
* Any active malignancy (other than non-melanoma skin cancer or localized cervical cancer or localized and presumed cured prostatic cancer) within the last 5 years with ongoing systemic treatment
* Cancer in contact with the internal and/or common carotid artery
* Extension of OPSCC across the midline of the base-of-tongue
* Arytenoid involvement in case of SGSCC
* Infiltration of apex for piriform sinus in case of HPSCC
* Cancer originating from the soft palate or posterior pharyngeal wall
* Requirement of a reconstruction with a free or regional flap (i.e. involvement of >50% of the soft palate)
* Pre-existing dysphagia not related to the oropharyngeal cancer or diagnostic biopsies
* Any psychological, cognitive, familial, sociological or geographical condition potentially hampering compliance with the study protocol, completion of patient reported measures and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the MD Anderson Dysphagia Inventory (MDADI) score | at 4.5 and 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Christian Simon, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (32):
- Belgium (4):
  - CHU-UCL Namur - CHU Mont Godinne, Namur, Yvoir
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet-Hopital Universitaire ULB, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Hopitaux Universitaires de Strasbourg - Hautepierre, Strasbourg, France
- Germany (9):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetklinikum Halle - Martin Luther Universitaet, Halle
  - Universitaets Krankenhaus Eppendorf - UKE - University Cancer Center, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Staedtisches Klinikum Leipzig - Klinikum St Georg, Leipzig
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Rechts der isar Der Technische Universitaet Muenchen, München
  - Universitaetsklinikum Tuebingen- Crona Kliniken, Tübingen
  - Universitaetsklinikum Ulm-Michelsberg-HNO, Ulm
- Italy (2):
  - Istituto Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia, Milan
- The Great Poland Cancer Centre, Poznan, Poland
- Spain (3):
  - Hospital Universitario Donostia, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - UniversitaetsSpital Zurich - Klinik fur Ohren, Hals und Gesichtschirurgie, Zurich
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - Cambridge University Hospital NHS - Addenbrookes Hospital, Cambridge
  - Cardiff and Vale University Health Board - University Hospital of Wales, Cardiff
  - Hull and East Yorkshire Hospitals NHS Trust - Castle Hill Hospital, Cottingham
  - Aintree University Hospital NHS Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation trust - Guy s and St Thomas' NHS - Guy's Hospital, London
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - South Tees Hospitals NHS Foundation Trust - The James Cook University Hospital, Middlesbrough